CLINICAL TRIAL: NCT06776068
Title: Comparison of the Impact of Lumboscopy and Laparoscopy on Ventilatory Mechanics in Patients Undergoing Nephrectomy
Brief Title: The Impact of Lumboscopy Versus Laparoscopy on Ventilatory Mechanics
Status: Not yet recruiting | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Roberto Gonzalez Cornejo, Anesthesiologist, University of Chile
Other Study IDs: CR/23053
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia; Mechanical Ventilation; Respiratory Physiology
Keywords: Anesthesia; Lumboscopy; Mechanical Ventilation; Laparoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients undergoing general anesthesia for laparoscopic and lumboscopic nephrectomy: Adult patients undergoing general anesthesia for laparoscopic and lumboscopic nephrectomy.

SUMMARY:
There are several techniques for performing minimally invasive urological surgeries. Among them, laparoscopic surgery, robotic surgery, and lumboscopy are noteworthy (1). The medical literature extensively documents the impact of pneumoperitoneum a procedure involving the insufflation of the peritoneal cavity with carbon dioxide (CO2), which is essential for laparoscopic and robotic surgeries on ventilatory mechanics.

As an alternative, CO2 insufflation into the retroperitoneum, as utilized in lumboscopic surgery, has been proposed. This approach is believed to exert a lesser impact on respiratory function and pulmonary mechanics. However, it is important to note that no conclusive evidence has yet been found to support this claim.

Assessing the impact of lumboscopic surgery could help establish it as a viable alternative for patients with pulmonary conditions, where mechanical ventilation poses significant challenges. To explore this possibility, a physiological study was designed to compare the effects of laparoscopic and lumboscopic surgery on ventilatory mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* ASA PS II-III
* Elective surgery
* Surgery: Partial or total nephrectomy

Exclusion Criteria:

* Severe pulmonary pathology
* Severe cardiovascular pathology
* Open surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing general anesthesia for minimally invasive nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Parameters of ventilatory mechanics | intraoperative
  Static compliance Plateau pressure Driving pressure Transpulmonary pressure

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Hospital Clínico Universidad de CHile, Santiago
  - Instituto Nacional del Cáncer, Santiago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guillonneau B, Ballanger P, Lugagne PM, Valla JS, Vallancien G. Laparoscopic versus lumboscopic nephrectomy. Eur Urol. 1996;29(3):288-91. doi: 10.1159/000473762. PMID 8740033